CLINICAL TRIAL: NCT03217526
Title: Investigation of the Effect of Different Gait Training on Physical Functions in Patients With Lower Extremity Burn Injury
Brief Title: Gait Training in Patients With Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, MsC, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GO 16/786
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-02

CONDITIONS: Burns; Gait Training; Physical Functions
Keywords: Burn injury; Gait; Physical Function
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ex Group (Active Comparator): EX: Standard exercise program (EX) (active range-of otion exercises, balance and mobility exercises) and walking training on the overground.
  This rehabilitation program physiotherapist will be applied to participants for five days a week. Walking training will be applied according to the gait speed determined by GAITRite computerized gait analysis system at initial assessment. Individuals will be instructed to walk with verbal commands and encourage them to continue their walk at constant speed.The duration of walking training will be recorded every day. The walking time will be determined according to the fatigue level of the individual. The level of fatigue of the individual will be questioned according to the modified borg scale.
  Interventions: Other: Gait Training
- Ex +WT Group (Experimental): Ex: A standard exercise (SE) (active range-of otion exercises, balance and mobility exercises) WT: walking training on the treadmill (WT). This rehabilitation program physiotherapist will be applied to participants for five days a week.Walking training will be applied according to the gait speed determined by GAITRite computerized gait analysis system at initial assessment. Individuals will be trained on the treadmill.The duration of walking training and the speed of walking training will be recorded every day. The walking time will be determined according to the fatigue level of the individual. The level of fatigue of the individual will be questioned according to the modified borg scale.
  Interventions: Other: Gait Training

INTERVENTIONS:
Other: Gait Training — Gait Training: Training will be applied by a physiotherapist on a treadmill or on an overgorund.

SUMMARY:
Twenty-four individuals with burn injury will be included in this study. Participants with burn injury will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass index; burn caharacteristics; type of burn injury, degree of burn injury, localization of burn injury and total burn surface area will be recorded. Gait parameters (step length, stride length, base support, step time, cycle time, cadence, velocity, single support, double support, swing ( % of gait cycle) and stance (% of gait cycle). will be recorded via GAITRite system.

DETAILED DESCRIPTION:
Twenty-four individuals with lower extremity burn injury will be included in this study. Participants will be included if they are aged of 18-50, able to walk independently at least 10 meters.

Participants will be divided in two groups; Intervention and control groups. Intervention group: standart rehabilitation program and gait training on the overground will be applied.

Conntrol Group:standart rehabilitation program and gait training on the treadmill will be applied.

Rehabilitation program will applied by physiotherapist during the acute hospitalization. Standart rehabilitation will include active range of motion exercises, functional mobility, balance activities.

Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass index; burn caharacteristics; type of burn injury, degree of burn injury, localization of burn injury and total burn surface area will be recorded. GAITRite system for gait parameters (step length, stride length, base support, step time, cycle time, cadence, velocity, single support, double support, swing ( % of gait cycle) and stance (% of gait cycle), timed up and go test (TUG) for dynamic balance and six minute walk test (6MWT) for exercise capacity, will be used. These evaluations will be made twice; initial (admission) and final (discharge).

ELIGIBILITY:
Inclusion Criteria:

* participiants who have lower extremity burn injury and able to walk independently 10 meters

Exclusion Criteria:

* f there is a medical condition that prevents the ambulance of the individual and oxygen is needed for ambulance, participants will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Cadence | It will be measured while walking on a GITRite system. It is about 5 meters electronically sensored carpet. Inıtially evaluation at first minute
  Walking speed
step length | Inıtially evaluation at first minute. It will be measured while walking on a GITRite system. It is about 5 meters electronically sensored carpet.
  Step Lenght assessment while walking

SECONDARY OUTCOMES:
six minute walk test | the distance at the en of Six minute
  this test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes The distance at the end of six minute will be recordedn.
Timed up and go test | Inıtially evaluation in first minute
  The patient sits in the chair with his/her back against the chair back On the command "go", the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down Timing begins at the instruction "go" and stops when the patient is seated. The time will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozkal O, Kismet K, Konan A, Hayran M, Topuz S. Treadmill versus overground gait training in patients with lower limb burn injury: A matched control study. Burns. 2022 Feb;48(1):51-58. doi: 10.1016/j.burns.2021.04.019. Epub 2021 Apr 24. PMID 34154896